CLINICAL TRIAL: NCT00262223
Title: Combined Treatment for Alcohol-Dependent Individuals With PTSD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Denise Hien, Principal Investigator, New York State Psychiatric Institute
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: #6266R-NIAAAHIE014341; R01AA014341-06 (NIH)
Record Dates: First submitted 2005-12-05; First posted 2005-12-06 (Estimated); Results first posted 2014-09-16 (Estimated); Last update posted 2020-03-03 (Actual); Status verified 2020-02

CONDITIONS: Stress Disorders, Post-Traumatic; Alcohol Abuse; Substance-Related Disorders
Keywords: Co-morbid alcohol dependence and PTSD; Alcohol and other drug use disorders; Treatment outcome
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Alcoholism; Substance-Related Disorders | interventions — Sertraline

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1) Seeking Safety + Sertraline (Active Comparator): Seeking Safety + Sertraline
  Interventions: Behavioral: Seeking Safety; Drug: Sertraline
- 2) Seeking Safety + Placebo (Placebo Comparator): Seeking Safety + Placebo;
  Interventions: Behavioral: Seeking Safety; Drug: Pill placebo

INTERVENTIONS:
Behavioral: Seeking Safety — Seeking Safety cognitive-behavioral treatment intervention for comorbid PTSD and substance use disorders
Drug: Sertraline — An anti-depressant medication, selective serotonin reuptake inhibitor (SSRI) type
  Other Names: Zoloft
  Arms: 1) Seeking Safety + Sertraline
Drug: Pill placebo
  Arms: 2) Seeking Safety + Placebo

SUMMARY:
This treatment intervention trial is designed for men and women with either alcohol misuse (e.g. hazardous or binge drinking) or alcohol use disorders (alcohol abuse or dependence) and comorbid PTSD. Participants will be randomly assigned to one of two treatments (a cognitive behavioral treatment intervention called "Seeking Safety" + Medication ("Zoloft") or Seeking Safety + placebo) and will be evaluated at baseline, at completion of the treatment (12 sessions over 12 weeks), and again at 6 months and 12 months post-treatment.

DETAILED DESCRIPTION:
The impetus for the current study is to contribute to the development of effective treatments targeted for men and women with either alcohol misuse (e.g., hazardous or binge drinking) or alcohol use disorders (e.g. alcohol abuse or alcohol dependence) and comorbid PTSD. Research findings have shown that these individuals have poorer treatment outcomes and show more severe symptoms than treatment seeking alcohol-misusing or alcohol dependent participants without PTSD. The aim of this study is to replicate and expand on 1) pilot studies demonstrating the effectiveness of a manualized cognitive-behavioral treatment specifically designed for individuals with comorbid substance use disorders and PTSD, "Seeking Safety" 2) preliminary results on the effectiveness of the antidepressant sertraline ("Zoloft") for a dually diagnosed population and 3) the examination of the effectiveness of these interventions over either treatment alone. We are comparing "Seeking Safety" alone to "Seeking Safety" in combination with the antidepressant medication sertraline ("Zoloft") in terms of their effectiveness in reducing alcohol use and PTSD symptoms. Participants will be randomly assigned to one of two treatments (Seeking Safety + Med or Seeking Safety + placebo) and will be evaluated at baseline, at completion of the treatment (12 sessions over 12 weeks), and again at 6 months and 12 months post-treatment. Secondary aims of the study include exploring potential differences between alcoholic subtypes on treatment outcomes; impact of combined treatment on treatment participation and global psychiatric symptoms; differences in the time course and order of changes in alcohol and drug use and PTSD symptoms by condition.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females who are a minimum of 18 years and maximum of 65 years.
2. Participants meet Diagnostic and Statistical Manual Diploma in Social Medicine IV (DSM-IV) criteria for current alcohol misuse, abuse or dependence.
3. Participants must have current alcohol use over past 90 days defined by more than or equal to 2 heavy drinking days or more than or equal to 14 drinks over 30 consecutive days or abstinence less than or equal to 21 consecutive days.
4. Participants meet criteria for full or subthreshold PTSD. Subthreshold PTSD criteria differs from full PTSD in that the individual meets cluster C (numbing) OR cluster D (hyperarousal) whereas full PTSD requires that the individual meets both cluster C and D.
5. Participants demonstrate no gross organic mental syndrome.
6. Participants are capable of giving informed consent and capable of complying with study procedures.
7. Participants speak English.

Exclusion Criteria:

1. Individuals who are at significant risk for suicide based on their current mental state or history.
2. Participants with other current Axis I psychiatric disorders that, in the investigators' judgment, are unstable and would be disrupted by study medications. Current diagnosis of Bipolar I and psychotic disorders are exclusionary.
3. Participants who are currently severely depressed.
4. Participants with a history of psychosis or mania.
5. Participants with organic mental syndrome.
6. Participants physiologically dependent on any substance other than alcohol (excluding nicotine or caffeine or medically stable and managed methadone).
7. Participants with comorbid substance abuse disorder who require detoxification treatment.
8. Participants with unstable or significant physical disorders (e.g., uncontrolled hypertension, poorly-controlled diabetes, alanine aminotransferase/aspartate aminotransaminase (AST/ALT) three times the upper limit of normal) that would increase the risk of study participation.
9. Participants with a known history of seizures (not related to alcohol withdrawal).
10. Participants with moderate to severe alcohol withdrawal that would require pharmacological intervention.
11. Participants currently taking prescribed psychotropic medication that is contraindicated for use with sertraline (e.g. antidepressant medications except for mirtazapine or trazodone when used for the treatment of insomnia ) and/or psychotropic medications where the participant has not achieved a stabilized regimen. Participants that are stable on medications that are not contraindicated with the use of sertraline (e.g., Methadone or Adderall) will not be excluded.
12. A history of an allergic reaction to sertraline.
13. Women who are currently pregnant or are trying to get pregnant or are nursing or are pre-menopausal and sexually active but not using effective birth control.
14. Participants refusing to be audio or videotaped.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2006-05; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Denise A. Hien, PhD, Principal Investigator — City College of New York & New York State Psychiatric Institute/Columbia University
Locations (1):
- City College, City University of New York, New York, New York, United States

REFERENCES:
- [Result] Hien DA, Levin FR, Ruglass LM, Lopez-Castro T, Papini S, Hu MC, Cohen LR, Herron A. Combining seeking safety with sertraline for PTSD and alcohol use disorders: A randomized controlled trial. J Consult Clin Psychol. 2015 Apr;83(2):359-69. doi: 10.1037/a0038719. Epub 2015 Jan 26. PMID 25622199
- [Result] Ruglass LM, Pedersen A, Cheref S, Hu MC, Hien DA. Racial differences in adherence and response to combined treatment for full and subthreshold post-traumatic stress disorder and alcohol use disorders: A secondary analysis. J Ethn Subst Abuse. 2016 Oct-Dec;15(4):434-448. doi: 10.1080/15332640.2015.1056927. Epub 2015 Sep 30. PMID 26422415

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants in the metropolitan New York area were recruited through newspaper and radio advertisements, flyers, and referrals from outpatient mental health centers between April 2006 and March 2012.
Pre-assignment Details: Individuals were screened through a brief telephone interview and then completed a baseline interview. After baseline assessment and medical clearance, eligible participants began a one-week, single-blind placebo lead-in phase. Those who completed the lead in phase were accepted into the study.
Groups:
- 2) Seeking Safety + Placebo: Seeking Safety + Placebo;
  Seeking Safety: Seeking Safety cognitive-behavioral treatment intervention for comorbid PTSD and substance use disorders
  Sertraline: An anti-depressant medication, selective serotonin reuptake inhibitor (SSRI) type
Period: Treatment Phase
Arm/Group | 1) Seeking Safety + Sertraline | 2) Seeking Safety + Placebo
Started | 32 | 37
Completed | 28 | 29
Not Completed | 4 | 8
Not completed — Withdrawal by Subject | 3 | 6
Not completed — Adverse Event | 1 | 2
Period: 1-week Post-treatment Follow-up
Arm/Group | 1) Seeking Safety + Sertraline | 2) Seeking Safety + Placebo
Started | 28 | 29
Completed | 24 | 25
Not Completed | 4 | 4
Not completed — Lost to Follow-up | 4 | 4
Period: 6-month Post-treatment Follow-up
Arm/Group | 1) Seeking Safety + Sertraline | 2) Seeking Safety + Placebo
Started | 28 (Subjects were included in subsequent follow-ups even if lost to contact during previous follow-up.) | 29 (Subjects were included in subsequent follow-ups even if lost to contact during previous follow-up.)
Completed | 22 | 28
Not Completed | 6 | 1
Not completed — Lost to Follow-up | 6 | 1
Period: 12-month Post-treatment Follow-up
Arm/Group | 1) Seeking Safety + Sertraline | 2) Seeking Safety + Placebo
Started | 28 (Subjects were included in subsequent follow-ups even if lost to contact during previous follow-up.) | 29 (Subjects were included in subsequent follow-ups even if lost to contact during previous follow-up.)
Completed | 21 | 22
Not Completed | 7 | 7
Not completed — Lost to Follow-up | 7 | 7

BASELINE CHARACTERISTICS:
Groups:
- 1) Seeking Safety + Sertraline: Seeking Safety, a cognitive-behavioral treatment intervention for comorbid PTSD and substance use disorders + Setraline, an anti-depressant medication, selective serotonin reuptake inhibitor (SSRI) type
- 2) Seeking Safety + Placebo: Seeking Safety, a cognitive-behavioral treatment intervention for comorbid PTSD and substance use disorders + Pill placebo
- Total: Total of all reporting groups
Arm/Group | 1) Seeking Safety + Sertraline | 2) Seeking Safety + Placebo | Total
Number analyzed (Participants) | 32 | 37 | 69
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.2 (9.8) | 42.5 (8.5) | 42.5 (9.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 30 | 56
  Male | 6 | 7 | 13

OUTCOME MEASURES:

1. Primary Outcome: Heavy Drinking Days/Week
Time Frame: Baseline, End-of-treatment, 6-month follow-up and 12-month follow-up
Measure: Mean (Standard Deviation); unit: Days/Week
Groups:
- 2) Seeking Safety + Placebo: Seeking Safety + Placebo
Arm/Group | 1) Seeking Safety + Sertraline | 2) Seeking Safety + Placebo
Number analyzed (Participants) | 32 | 37
Days/Week
  Baseline | 3.13 (2.17) | 2.89 (2.35)
  End-of-treatment | 1.05 (1.79) | 0.48 (1.69)
  6-month | .86 (1.46) | 0.75 (1.53)
  12-month | 0.30 (0.47) | 0.24 (0.44)
Statistical Analysis 1: Comparison: 1) Seeking Safety + Sertraline vs 2) Seeking Safety + Placebo; Between group analyses were conducted of time-by-treatment interaction that included the four study time points (baseline, end-of-treatment, 6-mos and 12-mos); Test type: Superiority or Other; p = 0.34, Generalized Estimating Equations; Negative binomial models with log link were applied to the alcohol consumption measure; Incidence Rate Ratio = 1.60, 95% CI 2-sided [0.61 to 4.23]

2. Primary Outcome: PTSD Symptom Severity / Clinician Administered PTSD Scale
Description: Clinician Administered PTSD Scale (CAPS) is a 17-item, semi-structured interview of PTSD symptoms. Range of scores is 0-136. Five rationally derived severity score ranges for interpreting CAPS total score have been proposed: 0-19 = asymptomatic/few symptoms, 20-39 = mild PTSD/subthreshold, 40-59 = moderate PTSD/threshold, 60-79 = severe PTSD symptomatology, and >80 = extreme PTSD symptomology (Weathers et. al., 2001). A 15-point change in CAPS total severity score has been proposed as a marker of clinically significant change (Weathers et. al., 2001).
Time Frame: Baseline, End-of-treatment, 6-month follow-up and 12-month follow-up
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 1) Seeking Safety + Sertraline | 2) Seeking Safety + Placebo
Number analyzed (Participants) | 32 | 37
units on a scale
  Baseline | 65.50 (20.03) | 59.50 (18.97)
  End-of-treatment | 36.25 (28.23) | 41.88 (29.30)
  6-month | 30.09 (20.70) | 37.46 (25.88)
  12-month | 24.90 (19.95) | 31.82 (24.44)
Statistical Analysis 1: Comparison: 1) Seeking Safety + Sertraline vs 2) Seeking Safety + Placebo; Generalized estimating equations (GEE) were utilized to model PTSD outcomes. This method is an extension of the generalized linear model that handles correlated data arising from repeated measurements, requires no parametric distribution assumption, and provides robust inference with respect to misspecification of the within-subject correlation. A temporal within-subjects autoregressive [AR(1)] correlation matrix was used to model participants across timepoints; Test type: Superiority or Other; p = 0.04, Generalized Estimating Equations — A trend-level time-by-treatment interaction (p = .096) was probed for simple effects, which revealed a significantly greater reduction in CAPS scores at end-of-treatment in the SS+Sertraline group relative to the SS+Placebo group; Parameter Estimate = -16.15, 95% CI 2-sided [-31.18 to -1.13]

ADVERSE EVENTS:
Groups:
- Seeking Safety + Sertraline: Seeking Safety, a cognitive-behavioral treatment intervention for comorbid PTSD and substance use disorders, + Setraline, an anti-depressant medication, selective serotonin reuptake inhibitor (SSRI) type
- Seeking Seeking + Placebo: Seeking Safety, a cognitive-behavioral treatment intervention for comorbid PTSD and substance use disorders + Pill Placebo
Arm/Group | Seeking Safety + Sertraline | Seeking Seeking + Placebo
Serious Adverse Events (participants affected / at risk) | 1/32 | 2/37
Other Adverse Events (participants affected / at risk) | 0/32 | 0/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Seeking Safety + Sertraline (N=32) | Seeking Seeking + Placebo (N=37)
Serious medical illness (General disorders) | 1 | 2 — Serious medical incidents were reported to the study's institutional review boards and none were determined to be study-related.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No